CLINICAL TRIAL: NCT05604664
Title: Clinical Value and Efficacy Index of Lymphadenectomy for Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Clinical Value and Efficacy Index of Lymphadenectomy for Thoracic Escc
Status: Completed | Type: Observational
Sponsor: Yongtao Han (Other)
Responsible Party: Sponsor-Investigator, Yongtao Han, Clinical Professor, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Other Study IDs: SCCH-TS2203
Record Dates: First submitted 2022-10-29; First posted 2022-11-03 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to to clarify the focus of lymph node dissection during esophagectomy.. The main question[s] it aims to answer is:

* provide a basis for accurate staging and the relationship between OS and lymph node dissection

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic findings proved ESCC (8th AJCC/UICC stage T1b-4aN0-3M0)
2. Underwent esophagecomy (two-field or three-field LN dissection)
3. The primary tumor was thoracic ESCC

Exclusion Criteria:

1. Located outside the thoracic
2. Patients underwent salvage or R1/R2 esophagecomy
3. The number of resected lymph nodes (RLNs) less than 15
4. With neoadjuvant therapy(NT) or salvage chemoradiotherapy(SCRT)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: (1) Pathologic findings proved esophageal cancer (8th AJCC/UICC stage T1b-4aN0-3M0). (2) underwent esophagecomy (two-field or three-field LN dissection). (3)The primary tumor was thoracic esophageal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1727 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
5-year survival rate of lymph nodes metastases (%) in patients | 2010.1.1-2017.12.30
  Surgical data were retrospectively collected

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided